CLINICAL TRIAL: NCT02500186
Title: The Clinical Study to Assess the Effect of the Amount of Carbohydrate Intake and Meals Differing in Glycemic Index (GI) in Patients Treated With a Sodium-dependent Glucose Cotransporter 2 (SGLT2) Inhibitor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kansai Electric Power Hospital (Other)
Collaborators: Medical Corporation Heishinkai OCROM Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kanden-hsp-0001; UMIN000017838 (Registry Identifier: UMIN)
Record Dates: First submitted 2015-07-02; First posted 2015-07-16 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Melltius, Type 2
MeSH Terms: interventions — 1,5-anhydro-1-(5-(4-ethoxybenzyl)-2-methoxy-4-methylphenyl)-1-thioglucitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- High GI meal containing 55% carbohydrate (Experimental): The energy intake of study patients is 1800 kcal per day. Study patients in high GI meal containing 55% carbohydrate group take 55% carbohydrate white rice diet.
  Interventions: Drug: Luseogliflozin; Other: Meal containing different carbohydrate ratio and GI value
- Low GI meal containing 55% carbohydrate (Experimental): The energy intake of study patients is 1800 kcal per day. Study patients in low GI meal containing 55% carbohydrate group take 55% carbohydrate brown rice diet
  Interventions: Drug: Luseogliflozin; Other: Meal containing different carbohydrate ratio and GI value
- High GI meal containing 40% carbohydrate (Experimental): The energy intake of study patients is 1800 kcal per day. Study patients in high GI meal containing 40% carbohydrate group take 40% carbohydrate white rice diet.
  Interventions: Drug: Luseogliflozin; Other: Meal containing different carbohydrate ratio and GI value

INTERVENTIONS:
Drug: Luseogliflozin — Study patients orally receive luseogliflozin 2.5 mg s.i.d. before breakfast for 7 days from the 8th day of starting the study meal to the 14th day.
  Other Names: Lusefi tab. 2.5mg
Other: Meal containing different carbohydrate ratio and GI value — High GI meal containing 55% carbohydrate Low GI meal containing 55% carbohydrate High GI meal containing 40% carbohydrate

SUMMARY:
The objectives of this clinical study is to assess the effect of the amount of carbohydrate intake and meals differing in glycemic index (GI) in patients of type 2 diabetes mellitus treated with an SGLT2 inhibitor (Luseogliflozin), which inhibits glucose reabsorption from renal uriniferous tubule, on glucose variability by using continuous glucose monitoring (CGM), and to establish dietary therapy which reduces the risk of hypoglycemia in patients treated with SGLT2 inhibitors. In addition, blood and urine samples are collected for metabolome analysis that will be performed as an extension study of the clinical study.

DETAILED DESCRIPTION:
<Background and Rationale> In order to decrease the risk of hypoglycemia caused by SGLT2 inhibitor, it is necessary to review the effect of the volume of carbohydrate intake and the level of GI value on variation of blood glucose.

Also, if a patient with chronic lack of carbohydrate intake receives SGLT2 inhibitors, there is a risk of serious hypoglycemic reaction. Thus, the establishment of proper meal for patients receiving SGLT2 inhibitors is the urgent task.

The objective of this study is to establish a safe dietary therapy for patients with type 2 diabetes mellitus to avoid hypoglycemia by controlling carbohydrate intake volume and GI value, where study patients are provided study meal three times a day and circadian blood glucose variation including blood glucose after meal is measured by using CGM.

In addition, blood and urine samples are collected for the future research (metabolome analysis) on the effect of carbohydrate intake volume and GI value on metabolism to be conducted as an extended study of this study.

<Study Procedures> Total of 24 study patients with type 2 diabetes mellitus who have not taken or washed out hypoglycemic drug (oral hypoglycemic drug and glucagon like peptide-1 receptor agonist) for at least 4 weeks are randomized into 3 groups (8 patients each) of high GI meal containing 55% carbohydrate group, low GI meal containing 55% carbohydrate group, and high GI meal containing 40% carbohydrate group. The energy intake of study patients in all the groups is 1800 kcal per day. Each study group patient takes the following diets for 14 days; study patients in high GI meal containing 55% carbohydrate group take 55% carbohydrate white rice diet; those in low GI meal containing 55% carbohydrate group take 55% carbohydrate brown rice diet; those in high GI meal containing 40% carbohydrate group take 40% carbohydrate white rice diet. Study patients orally receive luseogliflozin 2.5 mg s.i.d. before breakfast for 7 days from the 8th day of starting the study meal to the 14th day.

Planned examinations are conducted at the initiation of the study meal, the initiation of the study treatment, and the completion of the clinical study. Blood glucose is measured on 4 days from the 3rd day of the initiation of the study meal to pre-dose of study treatment and from 2 days before study treatment completion to the next day of study treatment so that blood glucose data of continuous 48 hours at one time can be obtained.

<Time and process of getting informed consents> Principal investigator or sub-investigator fully explains the clinical study to candidate patients using informed consent form approved by the Institutional Review Board prior to the study procedure and obtains written informed consent from subjects on voluntary basis after confirming that patients duly understand the content of the clinical study. Principal investigator or sub-investigator who gives explanation to patients and study patients affix a name and seal or give a signature and enter the date on the informed consent form. If study collaborator gives supplementary explanation, the collaborator also affixes a name and seal or give a signature and enter the date.

Principal investigator or sub-investigator provided the copy of the informed consent form to study patients who gave informed consent to participate in the clinical study and record them.

Principal investigator or sub-investigator documents the date of informed consent on case report form.

<Screening Examination> The eligibility for the clinical study of candidate patients who gave written informed consent are judged through the following examinations.

Candidate patients undergo screening examinations between 28 days and one day before the initiation of test meal (if the patient takes one hypoglycemic drug, between 28 days and one day before the initiation of washout).

Demographic background: date of birth, race, sex, disease duration of type 2 diabetes mellitus, drug and therapy used for treatment of type 2 diabetes mellitus within 3 months prior to the study procedure, complications / medical history, concomitant drug / therapy, drinking / smoking status, height / weight / BMI Examination item: physical examination, measurement of body fluid volume (by impedance method), clinical laboratory tests, vital signs (blood pressure, pulse rate, body temperature) <Statistical Analysis>

1. Demographic and Other Baseline Characteristics Efficacy analysis set and Safety analysis set are used for the analysis. For discrete values, frequency is summarized by group; for continuous data, summary statistics is calculated. Comparison between groups is also conducted.
2. Analysis of primary endpoint (Efficacy endpoint) Efficacy analysis set is used for the analysis. Summary statistics of blood glucose level by using CGM is calculated. Comparison between groups is also conducted.
3. Analysis of Secondary endpoint (Safety endpoint or efficacy endpoint) Safety analysis set and Efficacy analysis set are used for the analysis and the followings are summarized and analyzed.

   For discrete values of clinical laboratory tests and vital signs, frequency is summarized by group; for continuous data, summary statistics is calculated by group.

   Summary statistics of adverse event is calculated by group.
4. Significance level of test and confidence coefficient of confidence interval Tests are two-sided with the significance level of 5%. Confidence intervals are estimated with coefficient of 95%. <Sample size> Determination of sample size 24 patients (8 for each group) The sample size is 8 patients for each group because the size is operable and appropriate for analysis for the study.

<Action to be taken to study patients when an adverse event occurs> If an adverse event is observed, principal investigator or sub-investigator provides treatment or follow-up to the study patients until the patient recovers from the adverse event or the follow-up is judged to be unneccesary by medically explainable reason. If follow-up examination, additional examination, or re-examination is necessary, they are conducted after obtaining the study patient's informed consent.

Principal investigator or sub-investigator documents the name of adverse event, date of occurrence, intensity, seriousness, study drug adjustment, treatment for the adverse event, outcome, date of outcome, and relationship with the clinical study. For an adverse event which is observed from the initiation of the study drug administration to follow-up examination, the relationship with the study drug is also documented.

ELIGIBILITY:
Inclusion Criteria:

1. Japanese patients with type 2 diabetes
2. Patients aged 20 to 64, inclusive, when obtaining written informed consent, regardless of sex
3. Patients with HbA1c (NGSP) between 7.0 and 10.0 % at screening examination or patients with HbA1c (NGSP) <= 10.0 % (no lower limit) at screening examination if they receive one kind of hypoglycemic drug (oral hypoglycemic drug or GLP-1 receptor agonist)
4. Patients with BMI >= 20 kg/m2 and < 30 kg/m2
5. Outpatients
6. Patients who was explained about the clinical study, understood the content of the study, and gave written informed consent before participating in the clinical study

Exclusion Criteria:

1. Patients who are diagnosed as diabetes mellitus other than type 2 diabetes, e.g., type 1 diabetes, diabetes with specific mechanism or disease except for type 2 diabetes, pregnancy diabetes
2. Patients with complication of severe kidney dysfunction, e.g., nephrotic syndrome, renal failure, dialytic therapy
3. Patients with eGFR < 45mL/min/1.73m2 at screening examination
4. Patients with complication of severe hepatic disorder, e.g., hepatocirrhosis
5. Patients with complication of severe heart disease, e.g., cardiac infarction, cardiac failure, or of cerebral infarction, or patients with medical history of those within 6 months prior to the initiation of the clinical study (obtaining informed consent)
6. Patients who have serious complication of gastrointestinal disorders or who underwent a surgical operation that is known to affect the absorption of a drug by digestive tract
7. Patients with diabetic microangiopathy, e.g., retinopathy of diabetes, diabetic neuropathy, or others which cannot be fully controlled regardless of continuing treatment
8. Patients who are susceptible to dehydration (Patients with extremely poorly-controlled glycemia)
9. Patients with complication of malignancy (Patients who recovered from malignancy are permitted to participate in the clinical study)
10. Patients with a history of hypersensitivity to Luseogliflozin
11. Patients who is a chronic heavy drinker
12. Female patients who are pregnant, possibly pregnant, or breast-feeding
13. Other patients who are judged as ineligible for enrollment in the clinical study by the principal investigator or subinvestigat or subinvestigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose level using CGM | From Day 6 to Day 7, and from Day 13 and Day 14
  Early morning on 8th and 15th day after the initiation of test meal

SECONDARY OUTCOMES:
Change of Hematologic test (White blood cell) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Ratio of neutrophils) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Ratio of lymphocyte) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Ratio of monocyte) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Ratio of eosinophils) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Ratio of basophils) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Hemoglobin) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Hematocrit) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Hematologic test (Blood platelet) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Total cholesterol) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (High-density lipoprotein cholesterol) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Low-density lipoprotein cholesterol) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Triglyceride) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Albumin) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Total bilirubin) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Aspartate aminotransferase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Alanine aminotransferase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Lactase dehydrogenase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Alkaline phosphatase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (γ-glutamyltransferase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Creatine kinase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Amylase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Lipase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Blood urea nitrogen) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Urinary acid) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Lactic acid) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Ketone body) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Creatinine) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Natrium) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Kalium) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Chlorine) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Calcium) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Glucose) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Hemoglobin A1c) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Plasma fatty acid composition) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Non-esterified fatty acid) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Insulin) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (C-peptide) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Glucagon) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Choline esterase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Cross-linked N-telopeptide of type 1 collagen) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Biochemical examination of blood (Bone alkaline phosphatase) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary Qualitative (Sugar) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary Qualitative (Protein) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary Qualitative (Ketone body) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary Qualitative (Uric blood) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (Red blood cell) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (White blood cell) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (Squamous cell) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (Transitional cell) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (Urine creatinine) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (Urinary albumin) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Urinary sediment (Urinary cytology) from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Body temperature rate from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Blood pressure rate from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Change of Pulse rate from baseline (Day 1) to Day 15 | On Day 1 (before the start of test meal), Day 8 (pre-dose), and Day 15 (post-dose)
Adverse events | From screening examination to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Yutaka Seino, M.D., Ph.D., Study Director — Kansai Electric Power Hospital